CLINICAL TRIAL: NCT07268287
Title: Establishment of a Platform for the in Vivo Assessment of Therapies to Treat Metabolic Myopathies, Using Biomarkers and Stable Isotope Tracers to Evaluate Energy Metabolism: A First Step Towards Monitoring the Effectiveness of Innovative Therapies.
Brief Title: Assessment of Energy Metabolism in Metabolic Myopathies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Rajavel Elango, PhD, Principal Investigator, University of British Columbia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H20-01177
Record Dates: First submitted 2025-11-18; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Metabolic Myopathies
MeSH Terms: interventions — Urinalysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 13C-Glucose Breath Test (Experimental): Experiment piece 1:
  3 study days (pre-physio intervention) - single oral dose of unlabeled glucose and U-13C-glucose isotope.
  3 study days (post-physio intervention) - single oral dose of unlabeled glucose and U-13C-glucose isotope. Both in mg/kg/min.
  Interventions: Dietary Supplement: 13C-Glucose Breath Test
- Doubly Labelled Water & Urine Test (Experimental): Experiment piece 2:
  1 study day (pre-physio intervention) - single oral dose of doubly labelled water (2H218O) isotope.
  1 study days (post-physio intervention) - single oral dose of doubly labelled water (2H218O) isotope. Assess free-living total energy expenditure (in kcal).
  Interventions: Dietary Supplement: Doubly labelled water & urine test
- 12-week Physiotherapy Intervention (Experimental): Performed once by all participants, in between the pre- and post-intervention experiments described in the other arms.
  Interventions: Other: 12-week Physiotherapy Intervention
- Clinical Assessments - Exercise Test (Experimental): Experiment piece 3:
  1 study day (pre-intervention) and 1 study day (post-intervention).
  Exercise test: Maximum oxygen consumption (VO2 max) (in ml/kg/min).
  Interventions: Diagnostic Test: Clinical Assessments - Exercise Test
- Clinical Assessments - Muscle Content (Experimental): Experiment piece 3:
  1 study day (pre-intervention) and 1 study day (post-intervention).
  Muscle content test: Muscle mass measured by Dual-Energy X-ray Absorptiometry (DXA/DEXA) (in grams).
  Interventions: Diagnostic Test: Clinical Assessment - Muscle Content
- Clinical Assessments - Quality of Life Questionnaire (Experimental): Experiment piece 3:
  1 study day (pre-intervention) and 1 study day (post-intervention).
  Quality of life questionnaire test: Quality of life measure by pediatric quality of life questionnaire (PedsQL).
  Interventions: Diagnostic Test: Clinical Assessment - Quality of Life

INTERVENTIONS:
Other: 12-week Physiotherapy Intervention — A 12 week at-home physiotherapy exercises program performed at least 5 times per week, under virtual supervision 3 times per week by a kinesiologist, contains the same type of exercises that are normally prescribed to this population on a clinical basis. All patients will perform the same program to reduce inter-variability.
  Arms: 12-week Physiotherapy Intervention
Dietary Supplement: 13C-Glucose Breath Test — Experiment piece 1:
  Oral glucose isotope is administered to fasted participants on pre and post-intervention study days. Breath is collected over a 4-hour period following ingestion.
  Other Names:
  • D-glucose (Thermo Scientific™ NERL™ Trutol™)
  Arms: 13C-Glucose Breath Test
Dietary Supplement: Doubly labelled water & urine test — Experiment piece 2:
  1 study day pre and post-intervention fasted participants ingest a single oral dose of doubly labelled water (2H218O) isotope. 4 urine samples are collected over a 4 hour period following isotope administration, and once a day over 14 days.
  DLW is a safe and minimally invasive technique, considered the gold standard for precise measurement energy expenditure in humans. It involves enriching the body water with heavy hydrogen and oxygen (2H218O). The method is based on the principle that the 2H2 derived from body water is eliminated only as water (2H2O), while 18O is eliminated as both water (H2 18O) and carbon dioxide (C18O2).
  Arms: Doubly Labelled Water & Urine Test
Diagnostic Test: Clinical Assessments - Exercise Test — Experiment piece 3: Using a well-established clinical method VO2 max, once pre and post-intervention to assess for body composition (oxygen consumption during exercise).
  Arms: Clinical Assessments - Exercise Test
Diagnostic Test: Clinical Assessment - Muscle Content — Experiment piece 3: Using a well-established clinical method, DXA, once pre and post-intervention to assess for body muscle content (lean muscle mass)
  Arms: Clinical Assessments - Muscle Content
Diagnostic Test: Clinical Assessment - Quality of Life — Experiment piece 3: Using a well-established clinical survey, PedsQL, once pre and post-intervention to assess for participants perception of quality of life.
  Arms: Clinical Assessments - Quality of Life Questionnaire

SUMMARY:
Patients with metabolic myopathies suffer from exercise intolerance due to impaired ability to produce energy and secondary de-conditioning. There is a lack of methods enabling a non-invasive assessment of muscle energy production and studies regarding the benefits of therapeutic interventions are lacking as well. In this pilot study, the main aim is to assess the benefit of an intervention: a regular at home physiotherapy program for metabolic myopathies by measuring different outcomes pre and post therapeutic intervention using minimally invasive tests. The secondary aim of this study: investigators plan to describe the results of established non-invasive stable isotope tracer tests, namely, "glucose breath test" and "doubly labelled water & urine test" in patients pre and post 12 weeks at-home physiotherapy exercise program. The results of this study will be used for a larger scale study to assess energy metabolism in patients in patients with metabolic myopathies using non-invasive tests like breath and urine tests.

DETAILED DESCRIPTION:
Metabolic myopathies are a group of genetic conditions which affect the production of energy in the muscle and are caused by muscle adenosine triphosphate (ATP) depletion. This group includes disorders of mitochondrial oxidative phosphorylation (mitochondrial myopathies, MM), fatty acid oxidation (FAOD), Pompe disease and generation of glycolytic substrates (muscle glycogenosis, GSDs) from muscle glycogen. At large, these disorders are amenable to treatment including exercise and dietary treatment and/or vitamins cofactors supplementation.

There is a lack of non-invasive biomarkers which could be used to monitor treatment effectiveness. Traditionally, maximal oxygen consumption (VO2 max), quality of life questionnaire, dual-energy x-ray absorptiometry (DXA/DEXA), muscle biopsies, blood lactate and creatine kinase are used as a surrogate biomarker but have a limited validity to assess response to therapeutic interventions in patients with myopathies. The ultimate goal is to established a platform for clinical trials using minimally invasive tests to evaluate energy metabolism in patients with metabolic myopathies in response to therapeutic interventions, such as physiotherapy exercise program. These minimally invasive tests could be used to develop a platform for clinical trials for patients with muscle disease.

The main aim (objective) of this study is to assess the benefit of an intervention: a 12 weeks at-home physiotherapy exercises program for metabolic myopathies by measuring different outcomes pre and post therapeutic intervention using minimally-invasive tests. The investigators will administer a 12-week at-home physiotherapy exercises program to 3 metabolic myopathies pediatric patients between age 10 and 18 years.

The following outcomes will be measured pre and post intervention:

1. Glucose breath test: glucose oxidation (in mg/kg/min) measured by 13C glucose oxidation.
2. Doubly labelled water & urine test: assess free-living total energy expenditure (in kcal).
3. Exercise test: VO2 max (in ml/kg/min).
4. Muscle content test: Muscle mass (in grams) measured by DXA.
5. Quality of life questionnaire test: Quality of life measure by PedsQL.

The secondary aim (objective) of this study is to show that a glucose breath test measuring glucose oxidation (in mg/kg/min) and a doubly labelled water & urine test measuring total energy expenditure (in kcal) are outcomes that can be used in clinical trials to evaluate therapeutic interventions, along VO2 max, DXA and quality of life questionnaires. In that regard, this is a proof-of-concept study with the aim to describe the two biomarkers results in response to a therapeutic intervention in comparison to VO2-max and DXA scan and quality of life and clinical questionnaire in 3 participants.

The study design is n of 1 and will compare results of the tests pre and post therapeutic interventions in the same patients.

The glucose breath test: for the glucose oxidation (in mg/kg/min) measured by 13C glucose oxidation, results will be plotted as repeated measurements (3 times pre and post-intervention) for each individual participant. Repeat measurements will reduce the intra-individual variability. A 12 weeks at-home physiotherapy exercise protocol has been developed by the investigator team physician and kinesiologists experienced with exercise, children and metabolic myopathies. The therapeutic intervention, a 12 weeks at-home physiotherapy exercises program performed at least 5 times per week, under virtual supervision 3 times per week by a kinesiologist, contains the same type of exercises that are normally prescribed to this population on a clinical basis. All patients will perform the same program to reduce inter-variability.

In parallel, clinical methods such as VO2max, PedsQL and DXA will be measured pre- (baseline) and post-intervention evaluation. The investigators consulted a BCCHRI statistician with regard to the data analysis. Statistical analysis will include the intra-individual data analysis (n=1 study design) and will compare - using a Paired T test -the pre- and post- intervention data obtained from the two stable isotope tracer methods, VO2 max, DXA and quality of life questionnaires. The results of these tests will also be descriptively analyzed and the pre and post-intervention results will be plotted graphically.

The results of this proof of concept study will inform a larger scale project that was initially planned.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of the following: Mitochondrial Metabolic Myopathy (mMM), Fatty Acid Oxidation Disorder (FAOD), Pompe disease, or muscle Glycogen Storage Disease (GSD) (McArdle) via demonstration of deficient enzyme activity and / or demonstration of molecular testing confirming respective pathogenic variants and or compatible with disease phenotype.
* Age ≥10 years up to 18 years.
* Any gender.
* No past history of rhabdomyolysis requiring hospitalization.
* No signs or symptoms of infectious disease at least 14 days prior to the commencement of study visit (to mitigate the risk of rhabdomyolysis and coronavirus transmission).
* Participant must speak/understand English.
* Participant must have a smart phone or a tablet with a provider plan or that can be linked to Wi-Fi.
* Participant must have the time to commit to 11 visits at BC Children's Hospital over 21 weeks.

Exclusion Criteria:

* Any concurrent disorders / conditions that would interfere with /impact the study procedure (breath test and/or low intensity exercise).
* Diabetes Mellitus type I or II.
* Abnormal Cardiac assessment: cardiomyopathy or arrhythmia not allowing physical exercise.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2022-06-26 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2025-10-08 (Actual)

PRIMARY OUTCOMES:
Glucose Oxidation | 4 Hours
  Breath samples will be collected during the 3 pre and post-intervention study days to measure the rate of oxidation of 13C glucose (mg/kg/min).

SECONDARY OUTCOMES:
Doubly Labeled Water Free-living Total Energy Expenditure | 14 Days
  Energy expenditure can be calculated by measuring the difference in elimination rates of the heavy hydrogen and heavy oxygen in urine. The elimination rate is assessed from urine collected at the beginning and end of the observation period (~ 2 weeks). The 18O and 2H concentrations in urine are measured using isotope ratio mass spectrometry (IRMS). Assessed once pre- and post-intervention for free-living total energy expenditure (in kcal).
Clinical Assessments - Exercise Test | 1-2 Hours
  Exercise test: Maximal Oxygen Consumption (VO2 max) (ml/kg/min) during monitored exercise. Assessed once pre- and post-intervention.
Clinical Assessments - Muscle Content | 1 Hour
  Muscle content test: Lean muscle mass measured by Dual-Energy X-ray Absorptiometry (DXA/DEXA) (grams). Assessed once pre- and post-intervention.
Clinical Assessments - Quality of Life | 30 minutes
  Quality of life questionnaire test: Quality of life measure by the pediatric quality of life questionnaire (PedsQL) to assess for participants perceived mental, physical and emotional health. Assessed once pre- and post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Rajavel Elango, PhD, Principal Investigator — University of British Columbia; Catherine Brunel, MD, FRCPS, FCCMG, Principal Investigator — Provincial Health Services Authority British Columbia
Locations (1):
- BC Children's Hospital Research Institute, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided